CLINICAL TRIAL: NCT02644876
Title: Preventive Effects of Penehyclidine Hydrochloride Inhalation on Postoperative Pulmonary Complications in High-risk Patients: a Randomized, Double-blind, and Placebo Controlled Study
Brief Title: Preventive Effects of Penehyclidine Hydrochloride Inhalation on Postoperative Pulmonary Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015[06]; ChiCTR-IPC-15006603 (Registry Identifier: Chinese Clinical Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Complications
Keywords: Postoperative pulmonary complications; Selective anticholinergic bronchodilator; High risk patients; Postoperative period; Postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Injections; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penehyclidine group (Experimental): Penehyclidine inhalation will be administered (penehyclidine hydrochloride 0.5 mg/0.5 ml + normal saline 5.5 ml) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation will be performed with the high-flow oxygen-driven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Interventions: Drug: Penehyclidine inhalation
- Control group (Placebo Comparator): Placebo inhalation will be administered by inhalation (water for injection 0.5 ml + normal saline 5.5 ml ) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation will be performed with the high-flow oxygen-driven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Interventions: Drug: Placebo inhalation

INTERVENTIONS:
Drug: Penehyclidine inhalation — Penehyclidine inhalation will be administered by inhalation (penehyclidine hydrochloride 0.5 mg/0.5 ml, mixed with normal saline 5.5 ml) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation is performed with the high-flow oxygen-driven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Other Names: Penehyclidine Hydrochloride for Injection (Changtuoning)
  Arms: Penehyclidine group
Drug: Placebo inhalation — Placebo inhalation will be administered by inhalation (water for injection 0.5 ml, mixed with normal saline 5.5 ml) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation is performed with the high-flow oxygen-driven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Other Names: Water for injection
  Arms: Control group

SUMMARY:
Postoperative pulmonary complications (PPCs) are major causes of postoperative morbidity, mortality, and prolonged hospital stay.The incidence of PPCs may be as high as 41% to 75% in high-risk patients. Bronchodilator is frequently used in high-risk patients to prevent PPCs. Penehyclidine is a new anticholinergic agent which selectively block M1 and M3, but not M2 receptors. A pilot study of the investigators showed that prophylactic penehyclidine inhalation reduced the incidence of bronchospasm and the use of aminophylline in elderly patients after long-duration surgery. The purpose of this study is to investigate whether prophylactically penehyclidine inhalation could decrease the incidence of PPCs in high-risk patients after major intrathoracic and upper intraabdominal surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are major causes of postoperative morbidity, mortality, and prolonged hospital stay. The incidence of PPCs was found to vary from 2 to 19%, but this rate might be as high as 41 to 75% in patients after intrathoracic and intraabdominal surgery. According to Canet's model, the predicted incidence of PPCs in high-risk patients (ARISCAT risk index >= 45 points) is 42.1%. Use of effective strategies to prevent PPCs is essential for these patients.

Strategies that have been proved to be beneficial in decreasing PPCs include smoking cessation, proper management of chronic obstructive pulmonary disease before surgery, as well as use of lung-protective ventilation and goal-directed fluid therapy during surgery. Besides, bronchodilator inhalation is also helpful. Studies showed that, in high-risk patients undergoing intrathoracic surgery, airway resistance was increased due to bronchial hyperresponsiveness, which increased the risk of PPCs. Inhalation of anticholinergic bronchodilator can reduce the activity of vagus nerve and relieve high airway resistance, which may decrease the risk of bronchospasm and other PPCs.

It has been shown that M1, M3-receptor selective blockers have better effects than β2-receptor activator in dilating bronchia. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease (updated 2014) published by Global Initiative for Chronic Obstructive Lung Disease (GOLD) recommend the use of M1, M3-receptor selective blockers to relieve acute exacerbation of chronic obstructive pulmonary disease (COPD) and improve pulmonary function.

Penehyclidine hydrochloride is a new anticholinergic agent, which selectively blocks M1 and M3, but not M2 receptors. Preclinical studies found that it also has anti-inflammation effects. In a pilot study of the investigators, prophylactic inhalation of penehyclidine decreased the incidence of bronchospasm and the use of aminophylline in elderly patients after long-duration surgery. The investigators propose that prophylactic inhalation of penehyclidine might decrease the incidence of PPCs in high risk patients.

The purpose of this study is to investigate whether prophylactic penehyclidine inhalation could decrease the incidence of PPCs in high-risk patients after major intrathoracic and upper intraabdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age >50 years;
2. Scheduled to undergo upper abdominal or noncardiac thoracic surgery with expected duration ≥2 hours. For those who undergo laparoscopic or thoracoscopic surgery, the expected length of incision must be ≥5 cm;
3. Judged to be at high risk of PPCs according to the ARISCAT risk score (ARISCAT predictive score ≥45).

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical classification ≥IV or the expected survival duration ≤24 hours;
2. Preoperative history of symptomatic hypertrophy or glaucoma;
3. History of myocardial infarction, severe heart dysfunction (New York Heart Association functional classification ≥3) or tachyarrhythmia within one year;
4. Inhalation of β2-receptor activator, M-receptor blockers and/or glucocorticoids within one month before surgery;
5. Severe renal dysfunction (requirement of renal replacement therapy) or severe hepatic dysfunction (Child-Pugh grade C);
6. History of acute stroke within three months before surgery;
7. Refuse to participate in the study or unable to cooperate with the inhalation therapy;
8. Participation in other clinical trial during the last month or within the six half-life periods of the study drug used in the last trial.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications (PPCs) | Up to 30 days after surgery
  PPCs indicate complications that occur in the respiratory system from end of surgery till 30 days after surgery and require therapeutic intervention. Items include respiratory failure, respiratory infection, atelectasis, pleural effusion, bronchospasm, pneumothorax and aspiration pneumonitis.

SECONDARY OUTCOMES:
Time to onset of PPCs | From end of surgery till onset of first documented PPCs or death from any cause, whichever came first, assessed up to 30 days
  Time to onset of PPCs
Number of PPCs | Up to 30 days after surgery
  Items of PPCs include respiratory infection, atelectasis, pleural effusion, bronchospasm, respiratory failure, pneumothorax and aspiration pneumonitis.
Incidence of extrapulmonary complications | Up to 30 days after surgery
  Extrapulmonary complications indicate complications that occurred in the organs or systems other than the respiratory system and require therapeutic intervention.
Length of stay (LOS) in hospital after surgery | Up to 30 days after surgery
  Length of stay (LOS) in hospital after surgery
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hopital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Background] Brooks-Brunn JA. Predictors of postoperative pulmonary complications following abdominal surgery. Chest. 1997 Mar;111(3):564-71. doi: 10.1378/chest.111.3.564. PMID 9118688
- [Background] Thomsen T, Villebro N, Moller AM. Interventions for preoperative smoking cessation. Cochrane Database Syst Rev. 2014 Mar 27;2014(3):CD002294. doi: 10.1002/14651858.CD002294.pub4. PMID 24671929
- [Background] Kroenke K, Lawrence VA, Theroux JF, Tuley MR. Operative risk in patients with severe obstructive pulmonary disease. Arch Intern Med. 1992 May;152(5):967-71. PMID 1580723
- [Background] Celli BR. Perioperative respiratory care of the patient undergoing upper abdominal surgery. Clin Chest Med. 1993 Jun;14(2):253-61. PMID 8519171
- [Background] Hulzebos EH, Smit Y, Helders PP, van Meeteren NL. Preoperative physical therapy for elective cardiac surgery patients. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD010118. doi: 10.1002/14651858.CD010118.pub2. PMID 23152283
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Yan T, Wang D. [Effects of penehyclidine inhalation on postoperative pulmonary complications of elderly patients after long-duration surgery]. Zhonghua Yi Xue Za Zhi. 2014 Jan 14;94(2):122-6. Chinese. PMID 24721352
- [Background] Xiao HT, Liao Z, Tong RS. Penehyclidine hydrochloride: a potential drug for treating COPD by attenuating Toll-like receptors. Drug Des Devel Ther. 2012;6:317-22. doi: 10.2147/DDDT.S36555. Epub 2012 Nov 1. PMID 23139625
- [Background] Cui J, Li CS, He XH, Song YG. Protective effects of penehyclidine hydrochloride on acute lung injury caused by severe dichlorvos poisoning in swine. Chin Med J (Engl). 2013;126(24):4764-70. PMID 24342326
- [Background] Wu XJ, Xia ZY, Wang LL, Luo T, Zhan LY, Meng QT, Song XM. Effects of penehyclidine hydrochloride on pulmonary contusion from blunt chest trauma in rats. Injury. 2012 Feb;43(2):232-6. doi: 10.1016/j.injury.2011.10.009. Epub 2011 Nov 4. PMID 22055139
- [Background] Liu XB, Pan S, Yang XG, Li ZW, Sun QS, Zhao Z, Ma HC, Cui CR. Effect of penehyclidine hydrochloride on heart rate variability in hysteroscopy. Exp Ther Med. 2015 Jul;10(1):181-186. doi: 10.3892/etm.2015.2497. Epub 2015 May 18. PMID 26170932
- [Background] Wu GM, Mou M, Mo LQ, Liu L, Ren CH, Chen Y, Zhou J. Penehyclidine hydrochloride postconditioning on lipopolysaccharide-induced acute lung injury by inhibition of inflammatory factors in a rodent model. J Surg Res. 2015 May 1;195(1):219-27. doi: 10.1016/j.jss.2014.12.018. Epub 2014 Dec 17. PMID 25577143
- [Background] Ma TF, Zhou L, Wang Y, Qin SJ, Zhang Y, Hu B, Yan JZ, Ma X, Zhou CH, Gu SL. A selective M1 and M3 receptor antagonist, penehyclidine hydrochloride, prevents postischemic LTP: involvement of NMDA receptors. Synapse. 2013 Dec;67(12):865-74. doi: 10.1002/syn.21693. Epub 2013 Jul 24. PMID 23813456
- [Background] Shi H, Dong CM. [The effect of penehyclidine hydrochloride on the expression of inflammatory factor in rat with sepsis-associated lung injury]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2009 Nov;21(11):685-7. No abstract available. Chinese. PMID 19930890
- [Background] Xiao H, Liao Z, Meng X, Yan X, Chen S, Mo Z. Effects of the selective muscarinic receptor antagonist penehyclidine hydrochloride on the respiratory tract. Pharmazie. 2009 May;64(5):337-41. PMID 19530446
- [Background] Wang KW, Lin HQ, Wang JR. [Effect of penehyclidine hydrochloride as preoperation drug for elder on HRV]. Zhongguo Ying Yong Sheng Li Xue Za Zhi. 2008 Feb;24(1):28-9, 128. No abstract available. Chinese. PMID 21141550
- [Derived] Yan T, Liang XQ, Wang T, Li WO, Li HJ, Zhu SN, Wang DX. Prophylactic penehyclidine inhalation for prevention of postoperative pulmonary complications in high-risk patients: study protocol of a randomized controlled trial. Trials. 2017 Nov 28;18(1):571. doi: 10.1186/s13063-017-2315-7. PMID 29183393